CLINICAL TRIAL: NCT04248725
Title: Efficacy of a Telehealth Pain Self-Management Intervention in Employed Adults With Physical Disability: A Randomized Controlled Trial
Brief Title: Telehealth Pain Self-Management for Employed Adults
Acronym: E-TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dawn Ehde, Professor, School of Medicine: Rehabilitation Medicine:Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005686; A133507 (Other Grant/Funding Number: NIDILRR); 90RTEM0001-01-00 (Other Grant/Funding Number: ShirleyRyan Ability Lab)
Record Dates: First submitted 2020-01-08; First posted 2020-01-30 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Brain Injuries, Traumatic; Multiple Sclerosis; Spinal Cord Injuries; Amputation
Keywords: chronic pain; cognitive therapy; mindfulness meditation; activation skills; pain; employment; telehealth
MeSH Terms: conditions — Chronic Pain; Brain Injuries, Traumatic; Multiple Sclerosis; Spinal Cord Injuries; Pain

STUDY DESIGN:
Intervention Model Description: A randomized (1:1), single blind parallel-group trial comparing a telehealth pain self-management intervention, adapted to address employment issues (E-TIPS), to a waitlist control in adults with physical disabilities and chronic pain who are employed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-TIPS (Experimental): The E-TIPS intervention is based upon a cognitive-behavioral intervention for pain that was developed for and shown to be effective in people with chronic pain and a physical disability such as the conditions of interest in this study. Eight, 45-minute telephone sessions will be delivered by a clinician. A patient workbook will be used to facilitate skill acquisition and rehearsal in and outside of sessions. The intervention includes education about the role of unhelpful thoughts, particularly pain catastrophizing, and unhelpful pain coping behaviors; instruction in how to identify and change unhelpful or negative thinking about pain; utilization of helpful coping strategies; relaxation techniques; behavioral activation including setting goals for physical activation, activity pacing and scheduling; and coping with pain flare-ups. Each session includes a brief relaxation exercise. Participants receive digital audio recordings of relaxation exercises to practice at home.
  Interventions: Behavioral: E-TIPS
- Usual care (No Intervention): Participants assigned to the control intervention will continue to pursue standard care (a waitlist). Waitlist control subjects will be offered the opportunity to receive the intervention following completion of the final 6-month follow up outcome assessment.

INTERVENTIONS:
Behavioral: E-TIPS — Chronic pain self-management strategies for employed individuals with physical disabilities
  Arms: E-TIPS

SUMMARY:
The E-TIPS trial will evaluate an evidence-based, telehealth pain self-management intervention compared to standard care (a waitlist) for chronic pain in adults with physical disabilities who are employed. Participants from anywhere in the US will be randomized to either E-TIPS, a cognitive-behavioral pain self-management intervention delivered by telephone, or a waitlist control. Outcomes, including pain interference, will be assessed at baseline, mid-treatment, post-treatment, and 6-month follow up.

DETAILED DESCRIPTION:
Chronic pain is one of the most prevalent, disabling, and persistent comorbid conditions associated with physical disabilities, including limb loss, spinal cord injury, traumatic brain injury, and chronic neurodegenerative conditions such as multiple sclerosis. One half to two-thirds of adults with these conditions experience chronic pain. In addition to being associated with disability, depression, sleep disruption, and physical inactivity, chronic pain has deleterious social and societal costs, including job loss and reliance on long-term disability programs.

The E-TIPS intervention aims to address common barriers encountered by employed individuals with chronic pain. People with physical disabilities may be offered face-to-face delivery of pain self-management interventions, in clinical settings during business hours, which limits access to people with physical disabilities who are employed. These individuals must take time off work to attend multiple treatment sessions, overcome transportation difficulties, and contend with the stigma of seeking behavioral healthcare. Telehealth interventions, such as E-TIPS, have considerable potential for expanding the reach of pain self-management interventions for employed people with physical disabilities.

The proposed randomized (1:1), single-blind parallel-group trial will compare the E-TIPS telehealth pain self-management intervention to a waitlist control in adults with physical disabilities and chronic pain who are employed. Outcomes will be assessed before randomization, mid-treatment (6 weeks post-randomization), post-treatment (10 weeks post-randomization; primary endpoint), and 6-month follow up (25 weeks post-randomization). Participants will be recruited from across the US, including at University of Washington (UW) and Shirley Ryan AbilityLab (SRALab).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Self-reported physical disability
* Chronic pain defined as daily pain of ≥ 3 months duration and ≥ 3 average pain intensity in the past week on a 0-10 numerical rating scale
* Experiences pain for more than 45 out of the past 90 days (defined as 50% of the time or greater)
* Reads, speaks, and understands English
* Has access to and is able to communicate over the telephone with our without assistive devices
* Is employed, working 15-20 hours per week or more, on average, or earning in excess of substantial gainful activity (approximately $1200/month)

We will enroll individuals with a range of physical disabilities to maximize the generalizability of the results, because there is no evidence that the type of disability affects responsiveness to the proposed treatment

Exclusion Criteria:

* Under the age of 18
* Cannot read, speak, or understand English
* No self-reported physical disability
* Currently unemployed
* Plans to retire or leave employment within the study period
* Working fewer than 15-20 hours per week, on average, and earning less than approximately $1200 per month
* Cannot communicate or complete assessments over the phone or internet
* Chronic pain defined as daily pain of ≤ 3 months duration and ≤ 3 average pain intensity in the past week on a 0-10 numerical rating scale
* Experiences pain for fewer than 45 out of the past 90 days (defined as 50% of the time or less)
* Currently participating in another pain study or cognitive behavioral therapy (CBT) study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Ehde, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be deposited in a digital data repository. Direct and indirect identifiers will be removed to minimize disclosure risk. The data will be deposited with the digital repository of the Inter-university Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: on or or before October 1, 2024
Access Criteria: Data will be stored in a manner that enables retrieval and use at no cost to users. Each data set will use a Digital Object Identifier (DOI) for future reference and citation. Data submitted to ICPSR, will fit within the scope of the ICPSR Collection Development Policy found at this site: https://www.icpsr.umich.edu/icpsrweb/content/datamanagement/policies/colldev.html.
  ICPSR will make the research data from this project available to the broader social science research community. These files, in which direct and indirect identifiers have been removed to minimize disclosure risk, will be accessible directly through the ICPSR Web site. After agreeing to Terms of Use, users with an ICPSR MyData account may download the data at no cost.

REFERENCES:
- [Background] Ehde DM, Jensen MP, Engel JM, Turner JA, Hoffman AJ, Cardenas DD. Chronic pain secondary to disability: a review. Clin J Pain. 2003 Jan-Feb;19(1):3-17. doi: 10.1097/00002508-200301000-00002. PMID 12514452
- [Background] Dijkers M, Bryce T, Zanca J. Prevalence of chronic pain after traumatic spinal cord injury: a systematic review. J Rehabil Res Dev. 2009;46(1):13-29. PMID 19533517
- [Background] Ehde DM, Czerniecki JM, Smith DG, Campbell KM, Edwards WT, Jensen MP, Robinson LR. Chronic phantom sensations, phantom pain, residual limb pain, and other regional pain after lower limb amputation. Arch Phys Med Rehabil. 2000 Aug;81(8):1039-44. doi: 10.1053/apmr.2000.7583. PMID 10943752
- [Background] Krause JS, Cao Y, Clark JMR. Pain Intensity, Interference, and Medication Use After Spinal Cord Injury: Association With Risk of Mortality After Controlling for Socioeconomic and Other Health Factors. Arch Phys Med Rehabil. 2017 Dec;98(12):2464-2470. doi: 10.1016/j.apmr.2017.05.024. Epub 2017 Jun 23. PMID 28652067
- [Background] Negre-Pages L, Regragui W, Bouhassira D, Grandjean H, Rascol O; DoPaMiP Study Group. Chronic pain in Parkinson's disease: the cross-sectional French DoPaMiP survey. Mov Disord. 2008 Jul 30;23(10):1361-9. doi: 10.1002/mds.22142. PMID 18546344
- [Background] Franklin GM, Wickizer TM, Coe NB, Fulton-Kehoe D. Workers' compensation: poor quality health care and the growing disability problem in the United States. Am J Ind Med. 2015 Mar;58(3):245-51. doi: 10.1002/ajim.22399. Epub 2014 Oct 20. PMID 25331746
- [Background] Alschuler KN, Ehde DM, Jensen MP. The co-occurrence of pain and depression in adults with multiple sclerosis. Rehabil Psychol. 2013 May;58(2):217-21. doi: 10.1037/a0032008. PMID 23713732
- [Background] Kroenke K, Wu J, Bair MJ, Krebs EE, Damush TM, Tu W. Reciprocal relationship between pain and depression: a 12-month longitudinal analysis in primary care. J Pain. 2011 Sep;12(9):964-73. doi: 10.1016/j.jpain.2011.03.003. Epub 2011 Jun 16. PMID 21680251
- [Background] Anand P, Ben-Shalom Y. The promise of better economic outcomes for workers with musculoskeletal conditions. Roosevelt House: Public Policy Institute at Hunter College.2017.
- [Background] Social Security Administration. Annual Statistical Report on the Social Security Disability Insurance Program, 2015. Washington, DC2016.
- [Background] O'Connor AB, Schwid SR, Herrmann DN, Markman JD, Dworkin RH. Pain associated with multiple sclerosis: systematic review and proposed classification. Pain. 2008 Jul;137(1):96-111. doi: 10.1016/j.pain.2007.08.024. Epub 2007 Oct 24. PMID 17928147
- [Background] Warms CA, Turner JA, Marshall HM, Cardenas DD. Treatments for chronic pain associated with spinal cord injuries: many are tried, few are helpful. Clin J Pain. 2002 May-Jun;18(3):154-63. doi: 10.1097/00002508-200205000-00004. PMID 12048417
- [Background] Ehde DM, Dillworth TM, Turner JA. Cognitive-behavioral therapy for individuals with chronic pain: efficacy, innovations, and directions for research. Am Psychol. 2014 Feb-Mar;69(2):153-66. doi: 10.1037/a0035747. PMID 24547801
- [Background] Clarke G, Yarborough BJ. Evaluating the promise of health IT to enhance/expand the reach of mental health services. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):339-44. doi: 10.1016/j.genhosppsych.2013.03.013. Epub 2013 May 20. PMID 23701698

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 220 enrolled participants, 8 were excluded prior to the baseline assessment because they were not able to be contacted for baseline completion. After 212 enrolled participants completed the baseline assessment, 10 additional participants were excluded because: we were unable to contact them for randomization (n=5), they withdrew from the study due to personal circumstances (n=3), or withdrawn by staff (n=2). A total of 202 were randomized to one of the two study arms.
Period: Post-Treatment
Arm/Group | E-TIPS | Usual Care
Started | 102 | 100
Completed | 96 | 95
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5
Period: 6-Month Follow Up
Arm/Group | E-TIPS | Usual Care
Started (participants who did not complete Period 1's outcome assessment were offered the opportunity to complete Period 2's outcome assessment. Thus, 102 and 100, respectively, are correct for the numbers that started Period 2.) | 102 | 100 (see comment for ETIPS arm.)
Completed | 93 | 92
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-TIPS | Usual Care | Total
Number analyzed (Participants) | 102 | 100 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12) | 46 (12) | 46 (12)
Sex/Gender, Customized [Number; unit: participants]
  Female | 71 | 70 | 141
  Male | 31 | 30 | 61
  Man | 30 | 30 | 60
  Woman | 69 | 65 | 134
  Non-binary | 2 | 2 | 4
  Other | 0 | 1 | 1
  Prefer not to answer/unknown | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 88 | 88 | 176
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 12 | 17
  White | 80 | 71 | 151
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 102 | 100 | 202
Disability condition [Count of Participants; unit: Participants]
  Multiple sclerosis | 48 | 48 | 96
  Spinal cord injury | 17 | 20 | 37
  Traumatic brain injury | 13 | 12 | 25
  Amputation | 11 | 7 | 18
  Multiple diagnoses | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Interference
Description: Patient-reported pain interference using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale-6-item. Each item is scored 1 (not at all) to 5 (very much), yielding a raw score between 6 and 30, which is converted to a standard t-score. The population mean is a score of 50, with a standard deviation of 10. Higher scores indicate greater self-reported pain interference.
Time Frame: Baseline (week 0) and 12 weeks (post-treatment)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | E-TIPS | Usual Care
Number analyzed (Participants) | 102 | 100
T-score | -4.0 [-8.5 to 0.1] | -1.3 [-5.0 to 2.0]
Statistical Analysis 1: Comparison: E-TIPS vs Usual Care; Test type: Superiority; p = 0.004, Mixed Models Analysis; Models were adjusted for sex, baseline severity, and disability condition; Mean Difference (Net) = -2.7

2. Secondary Outcome: Change in Pain Self-efficacy
Description: Patient-reported pain self-efficacy for managing pain using the University of Washington Pain Self-Efficacy Scale-6 item. Each item is scored 1 (not at all) to 5 (very much), yielding a raw score between 6 and 30, which is converted to a standard t-score.The population mean is a score of 50, with a standard deviation of 10. Higher scores indicate greater patient-reported self-efficacy for managing pain.
Time Frame: Baseline (week 0) and 12 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | E-TIPS | Usual Care
Number analyzed (Participants) | 102 | 100
T-score | 5.5 (8.2) | 0.9 (7.5)
Statistical Analysis 1: Comparison: E-TIPS vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.59, 95% CI 2-sided [0.30 to 0.88]

3. Secondary Outcome: Change in Average Pain Intensity
Description: 0-10 Numerical Pain Rating Scale of average pain intensity in past week (0 = no pain, 10 = worst pain imaginable). Higher scores indicate higher levels of self-reported pain intensity; range of 0 - 10.
Time Frame: Baseline (week 0) and 12 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E-TIPS | Usual Care
Number analyzed (Participants) | 102 | 100
units on a scale | -0.9 (1.9) | -0.3 (1.7)
Statistical Analysis 1: Comparison: E-TIPS vs Usual Care; Test type: Superiority; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.61 to -0.03]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were identified during intervention sessions and assessments.
Arm/Group | E-TIPS | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/102 | 0/100
Other Adverse Events (participants affected / at risk) | 0/102 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-TIPS (N=102) | Usual Care (N=100)
Strained muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — While practicing progressive muscle relaxation, a participant overdid it and strained a muscle, leading to a temporary increase in pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT04248725/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT04248725/SAP_001.pdf